CLINICAL TRIAL: NCT02677480
Title: The Effect of Probiotic Streptococci and pH-rising Components on the Oral Microbial Flora in Subjects With Reduced Salivary Secretion Rate
Brief Title: The Effect of Probiotic Streptococci and pH-rising Components on the Oral Microbial Flora
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vinnova (Other Government); Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 662-08
Record Dates: First submitted 2015-11-19; First posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Hyposalivation
Keywords: Microflora; Probiotics; Hyposalivation; Lactobacilli; Mutans streptococci; pH-rising components
MeSH Terms: conditions — Xerostomia | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test group, probiotic tablets and gel (Active Comparator): Test group, probiotic tablets and gel: tablets with probiotic bacteria (10exp8/tablet) and pH-rising components and gel (with probiotic bacteria and pH-rising components) in trays on the teeth once a week.
  Interventions: Dietary Supplement: Test group, probiotic tablets and gel
- Placebo group, placebo tablets and gel (Placebo Comparator): Placebo group, placebo tablets and gel: placebo tablets without probiotic bacteria and pH-rising components and gel (with no probiotic bacteria but with pH-rising components) in trays on the teeth once a week.
  Interventions: Dietary Supplement: Placebo group, placebo tablets and gel

INTERVENTIONS:
Dietary Supplement: Test group, probiotic tablets and gel — Effect of probiotic tablets and gel on acidogenic bacteria
  Arms: Test group, probiotic tablets and gel
Dietary Supplement: Placebo group, placebo tablets and gel — Effect of placebo tablets and gel on acidogenic bacteria
  Arms: Placebo group, placebo tablets and gel

SUMMARY:
The test group consisted of eighteen subjects with hyposalivation used probiotic tablets (≥ 4/day) and gel (once a week) (streptococci, bicarbonate and carbamide) for 3 months and 9 used placebo tablets and gel. The salivary secretion rates were measured and microbial samples collected and analysed using cultivation technique twice both at baseline and at the 3-month follow up (1-2 weeks between the appointments).

DETAILED DESCRIPTION:
The aim was to analyse the effect of daily intake of probiotic alpha-haemolytic facultative anaerobic streptococci (Streptococcus oralis), pH-rising components and Stevia on the oral microflora in hyposalivated subjects.

Material and methods: Subjects with hyposalivation (unstimulated secretion rate of < 0.1 ml/min and/or a stimulated secretion rate < 0.7 ml/min) and ≥ 10 000 cfu/ml of mutans streptococci and/or lactobacilli on the tongue or in the supragingival plaque were included. Eighteen subjects used probiotic tablets (≥ 4/day) and gel (once a week) for 3 months and 9 used placebo tablets and gel. The salivary secretion rates were measured and microbial samples collected and analysed using cultivation technique twice both at baseline and at the 3-month follow up (1-2 weeks between the appointments).

ELIGIBILITY:
Inclusion Criteria:

* No open wounds in the oral cavity
* ≥ 10 own teeth
* Experienced dry mouth for at least 1 year
* An unstimulated salivary secretion rate < 0.1 ml/min
* A stimulated secretion rate < 0.7 ml/min and high numbers (≥ 10000 cfu/ml) of lactobacilli and/or mutans streptococci on the tongue and/or in dental plaque

Exclusion Criteria:

* Removable prosthesis
* Reduced immune defence
* Serious heart diseases
* Implanted joints or heart valves
* Lactose intolerance (the probiotic streptococci are freeze-dried in skim milk)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Reduction of proportions of mutans streptococci and/or lactobacilli in supragingival plaque and/or on the tongue at 3 months compared with baseline | 3 months
  The oral microflora of patients with hyposalivation (unstimulated secretion rate ≤ 0.1 ml/min and/or a stimulated secretion rate ≤ 0.7 ml/min) is analysed. Samples are collected from supragingival plaque and from the tongue and are analysed using cultivation techniques. The total microbial count is registered as well as numbers of streptococci, mutans streptococci and lactobacilli. Patients with counts of mutans streptococci and/or lactobacilli ≥ 10000 colony forming units/ml are randomly included in either the test group or in the placebo group. After 3 months, microbial samples are collected again from supragingival plaque and from the tongue and proportions of microorganisms analysed. Statistically significant differences in proportions of mutans streptococci and lactobacilli between baseline and after 3 months will be analysed using Students' paired t-test.

SECONDARY OUTCOMES:
Reduction of numbers of mutans streptococci and/or lactobacilli in supragingival plaque and/or on the tongue at 3 months compared with baseline | 3 months
  The oral microflora of patients with hyposalivation (unstimulated secretion rate ≤ 0.1 ml/min and/or a stimulated secretion rate ≤ 0.7 ml/min) is analysed. Samples are collected from supragingival plaque and from the tongue and are analysed using cultivation techniques. The total microbial count is registered as well as numbers of streptococci, mutans streptococci and lactobacilli. Patients with counts of mutans streptococci and/or lactobacilli ≥ 10000 colony forming units/ml are randomly included in either the test group or in the placebo group. After 3 months, microbial samples are collected again from supragingival plaque and from the tongue and the numbers of microorganisms analysed. Statistically significant differences in numbers of mutans streptococci and lactobacilli between baseline and after 3 months will be analysed using Students' paired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Annica Almstahl, Assoc. prof., Principal Investigator — Goteborg University
Locations (1):
- Institute of odontology, Gothenburg, Sweden